CLINICAL TRIAL: NCT02292732
Title: A Phase I, Open-Label Study to Determine the Effect of Repeat Dosing of Trametinib on the Pharmacokinetics and Safety of a Combined Oral Contraceptive (Norethindrone Plus Ethinyl Estradiol) and to Characterize the Pharmacokinetics of Trametinib's Metabolite M5 in Female Subjects With Solid Tumors
Brief Title: A Pharmacokinetics (PK) and Safety Study to Determine the Effect of Repeat Dosing of Trametinib on Combined Oral Contraceptive (Norethindrone Plus Ethinyl Estradiol) in Female Subjects With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113707
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: Pharmacokinetics; Solid Tumors; Safety; Trametinib; MEK Inhibitor; Combined Oral Contraceptive; Trametinib's Metabolite M5; Norethindrone; Ethinyl Estradiol
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trametinib/ ORTHO-NOVUM® tablet (Experimental): Subjects in treatment period 1will take one active tablet from the ORTHO-NOVUM® tablet 1/35 dial-pack once daily at approximately the same time each day for 21 days (Days 1 through 21), followed by one placebo tablet once daily at approximately the same time each day for 7 days (Days 22 through 28). In addition, subjects will take trametinib 2 mg (1 tablet) once daily at approximately the same time each day for a total of 17 days (Days 12 through 28). Subjects in treatment period 2 will take one active tablet from the ORTHO-NOVUM® tablet 1/35 dial-pack once daily at approximately the same time each day for 11 days (Days 1 through 11). In addition, subjects will take trametinib 2 mg (1 tablet) once daily at approximately the same time each day for 11 days (Days 1 through 11).
  Interventions: Drug: Trametinib 0.5 mg; Drug: Trametinib 2 mg; Drug: ORTHO-NOVUM® tablet 1/35; Drug: Placebo

INTERVENTIONS:
Drug: Trametinib 0.5 mg — Each tablet will contain GSK1120212B equivalent to 0.5 mg of Trametinib. Tablets are yellow, oval, biconvex, film-coated (4.85 x 8.86 millimeter [mm]) to be taken orally and once daily
Drug: Trametinib 2 mg — Each tablet will contain GSK1120212B equivalent to 2 mg Trametinib. Tablets are pink, round, biconvex and film-coated tablets (7.5 mm in diameter) to be taken orally and once daily.
Drug: ORTHO-NOVUM® tablet 1/35 — Each peach tablet will contain 1 mg of NE and 0.035 mg of EE. Other inactive ingredients will include lactose, magnesium stearate and pregelatinized corn starch
Drug: Placebo — Each green tablet will contain only inert ingredients: D&C yellow No. 10 Aluminum Lake, FD&C Blue No. 2 Aluminum Lake, lactose, magnesium stearate, microcrystalline cellulose, and pregelatinized cornstarch. The tablets are to be taken orally and once daily

SUMMARY:
This is a Phase I, open-label, non-randomized, sequential, two-period, repeat-dose study to evaluate the effect of trametinib 2 milligram (mg) once daily on the repeat-dose pharmacokinetic (PK) of an oral contraceptive (OC) containing norethindrone (NE) and ethinyl estradiol (EE) (ORTHO-NOVUM® tablets: 1 mg NE + 0.035 mg EE) in female subjects with solid tumors.

The study will determine PK interaction between trametinib and the components of combination oral contraceptives that would compromise the effectiveness of the contraceptives.

The study will also evaluate the repeat dose PK of trametinib and its metabolite M5 using a validated assay.

The study will enroll approximately 24 subjects. Each subject will participate in the study for approximately up to 13 to 15 weeks which will consist of a 30 day screening period, followed by 2 treatment periods (Period 1: 28 days and Period 2: ranging from 12 days to up to 21 days), and a transition visit or post-treatment follow-up visit. In Period 1, subjects will take one active tablet from the ORTHO-NOVUM® tablet 1/35 dial-pack once daily at approximately the same time each day for 21 days (Days 1 through 21), followed by one inert (referred to as placebo) tablet once daily at approximately the same time each day for 7 days (Days 22 through 28). In addition, subjects will take trametinib 2 mg (1 tablet) once daily at approximately the same time each day for a total of 17 days (Days 12 through 28). In Period 2, subjects will take one active tablet from the ORTHO-NOVUM® tablet 1/35 dial-pack once daily at approximately the same time each day for 11 days (Days 1 through 11). In addition, subjects will continue taking trametinib 2 mg (1 tablet) once daily at approximately the same time each day for 11 days (Days 1 through 11). ORTHO-NOVUM® is a registered trademark of Ortho Pharmaceutical Corporation.

ELIGIBILITY:
Inclusion Criteria:

* Is a female subject >=18 years but <59 years of age at the time of signing the informed consent.
* Has a histologically or cytologically confirmed diagnosis of a solid tumor malignancy (except for any excluded malignancies listed in Exclusion Criteria) that is not responsive to standard therapy(ies) or for which there is no approved therapy.
* Is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has a body mass index (BMI) within the range of 19 to 40 kilogram/squared meter (kg/m^2) (inclusive)
* Is a non-smoker or is willing to abstain from use of tobacco and/or nicotine-containing products from time of Screening until the post-treatment follow-up visit or transition to MEK rollover study (MEK114375).
* Meets one of the following criteria: Is currently on a stable regimen of ORTHO-NOVUM® tablet 1/35, or Is willing to switch to a regimen of ORTHO-NOVUM® tablet 1/35 from a stable regimen of an alternate OC, or Is willing to start a regimen of ORTHO-NOVUM® tablet 1/35
* Has a negative serum beta-human chorionic gonadotropin (Beta-hCG) pregnancy test within 7 days of first dose of study treatment
* Meets one of the following criteria: Is of non-childbearing potential - defined as females with a documented bilateral tubal ligation or tubal occlusion or hysterectomy without oophorectomy (at least one functioning ovary required); Is of childbearing potential and agrees to use an appropriate method of contraception in addition to the OC provided for at least 14 days prior to the first dose of study treatment until completion of the post-treatment follow-up visit or transition to the Mitogen-activated extracellular signal-regulated kinase (MEK) rollover study (MEK114375)
* Has no prior treatment- related toxicities >Grade 1 (except alopecia) at the time of enrollment
* Is able to swallow and retain orally administered medication
* Has adequate baseline organ function as follows: Hematologic (Absolute neutrophil count >=1.2 × 10^9/L; Hemoglobin >=9 g/dL; Platelets >=75 × 10^9/L; prothrombin time/international normalized ratio [PT/INR] and partial thromboplastin time [PTT] <=1.5x upper limit of normal [ULN]) ; Hepatic (Albumin >=2.5 g/dL; Total bilirubin <=1.5xULN [isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%]); alanine aminotransferase (ALT) <=2.5xULN; ALT with documented liver metastases or tumor infiltration; >2.5xULN but <=5xULN) ; Renal (Creatinine or <=1.5 ULN; Calculated creatinine clearance [calculated by the Cockcroft-Gault formula] >=50 milliliters/minute [mL/min]) ; Cardiac (left ventricular ejection fraction [LVEF] >= lower limit of normal [LLN] by echocardiogram [ECHO] or Multigated acquisition scan [MUGA])

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Had prior exposure to a MEK inhibitor
* Has one of the following excluded tumor types as trametinib therapy has been shown to have minimal benefit in these populations: BRAF V600E mutant melanoma and failed prior BRAF inhibitor therapy; Metastatic pancreatic cancer
* Has had any major surgery extensive radiotherapy, or anti-cancer therapy (e.g., chemotherapy with delayed toxicity, biologic therapy, or immunotherapy) within 21 days prior to enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrollment. Prolonged immobilization must have resolved prior to start of study.
* Has a known or suspected carcinoma listed below that is excluded as administration of ORTHO-NOVUM® tablet would be contraindicated: carcinoma of the breast, or carcinoma of the endometrium, or BRCA+ ovarian cancer, or other known or suspected estrogen-dependent neoplasia, or hepatocellular carcinoma
* Has a history of another malignancy: Exception: A subject who: has been disease-free for 3 years, or; has a history of completely resected non-melanoma skin cancer, or; has an indolent second malignancy, other than any of the excluded malignancies listed in the previous exclusion Criteria.
* Has a life expectancy of <3 months
* Has a history of interstitial lung disease or pneumonitis.
* Has a history of Retinal vein occlusion (RVO)
* Has a history of any of the following conditions that would contraindicate administration of an Oral contraceptive (OC): Uncontrolled or treatment refractory hypertension. NOTE: Treatment-refractory hypertension is defined as a blood pressure of systolic >140 millimeters of mercury (mmHg) and/or diastolic >90 mmHg which cannot be controlled by anti-hypertensive therapy; Diabetes mellitus (type 1 and 2) with vascular involvement (neuropathy./retinopathy/nephropathy); Stroke; Acute or past history of venous thromboembolism or known thrombophilia including factor V Leiden mutation; prothrombin mutation; protein S, protein C, and antithrombin deficiencies; or antiphospholipid antibodies; Migraine headaches (headaches with focal neurological symptoms); Undiagnosed abnormal uterine bleeding
* Has a Bazett-corrected QT (QTcB) interval >=480 milliseconds (msec) at Screening
* Has a LVEF, as measured by ECHO (preferred) or MUGA scan, below the institutional LLN, or if a LLN does not exist at an institution, <50%
* Has a history or current evidence of cardiovascular risk including any of the following: History or evidence of current clinically significant uncontrolled arrhythmias. NOTE: Subjects with controlled atrial fibrillation for >30 days prior to enrollment are eligible. History or evidence of current acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrolment. History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); Has an intra-cardiac defibrillator
* Has symptomatic or untreated leptomeningeal, brain metastases, or spinal cord compression. Note: Subjects previously treated for these conditions that have had stable central nervous system disease (verified with consecutive imaging studies) for >3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose of corticosteroids for at least 30 days prior to Day 1 are permitted.
* Has any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Is pregnant, lactating or actively breastfeeding.
* Is currently receiving a prohibited medication(s) or requires the use of any of the prohibited medication(s) during the study. NOTE: Use of anticoagulants such as warfarin is permitted; however, INR must be monitored in accordance with local institutional practice.
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody at Screening or within 3 months prior to first dose of study treatment . NOTE: Subjects with laboratory evidence of cleared hepatitis B virus and hepatitis C virus infection will be permitted.
* Has current or chronic history of liver disease or known hepatic or biliary abnormality (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment ). NOTE: Stable chronic liver disease defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice.
* Has participated in a clinical trial and received investigational drug(s) within 30 days, 5 half-lives or twice the duration of the biological effect of trametinib whichever is longer, prior to enrollment in this study.
* Has participated in a study that resulted in or made a donation of blood or blood products in excess of 500 mL within 56 days of the first dose of study treatment.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study treatment, or excipients.
* Has any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures

Ages: 18 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Composite of steady state PK parameters of NE and EE | Day 11 and Day 12 of both the treatment periods
  Steady state PK parameters will include Area under the concentration-time curve over the dosing interval (AUC[0-tau]), Maximum observed plasma concentration (Cmax), Pre-dose concentration (C0) and Time to Cmax (Tmax)
Composite of steady state PK parameters of NE and EE in combination with trametinib | Day 11 and Day 12 of both the treatment periods
  Steady state PK parameters will include AUC(0-tau), Cmax, C0 and Tmax

SECONDARY OUTCOMES:
Composite of steady state PK parameters of Plasma trametinib and M5 | Day 11 and Day 12 of treatment period 2
  Steady-state PK parameters will include AUC(0-tau), Cmax, C0, Tmax, and metabolite/parent AUC ratio
Safety and tolerability as assessed by measuring vital signs | Up to 107 days
  Vital signs will include measurement of blood pressure, temperature and pulse rate
Safety and tolerability as assessed by measuring electrocardiogram (ECGs) | Up to 107 days
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and Corrected QT interval (QTc) intervals. Electrocardiograms (ECGs) will be performed by qualified site personnel after the subject has rested at least 5 minutes in a semi-recumbent or supine position.
Safety and tolerability by assessing ECHOs | Up to 107 days
  The evaluation of the echocardiographer will include an evaluation for Left ventricular ejection fraction (LVEF) and both right and left-sided valvular lesions
Safety and tolerability by assessing clinical laboratory tests | Up to 107 days
  Clinical laboratory tests will include hematology, clinical chemistry, urinalysis and additional parameters
Safety and tolerability by assessing adverse events (AEs) | Up to 107 days
  AEs will be collected throughout the treatment periods up to follow up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline